CLINICAL TRIAL: NCT07247877
Title: Innovative Technology Research on Using Small-for-size Grafts for Auxiliary Liver Transplantation in the Treatment of Portal Hypertension
Brief Title: Research on Using Small-for-size Grafts for Auxiliary Liver Transplantation in the Treatment of Portal Hypertension
Status: Enrolling by invitation | Type: Observational
Sponsor: Ru-zhou Cai (Other)
Responsible Party: Sponsor-Investigator, Ru-zhou Cai, Principal Investigator, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: BFHHZML20250022
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- auxiliary liver transplantation using small-for-size grafts
- conventional liver transplantation using Standard-size graft

SUMMARY:
The objective of this observational study is to compare the safety profile of auxiliary liver transplantation using small-for-size grafts with that of conventional liver transplantation and to evaluate the efficacy of this technique. The primary research question it seeks to investigate is:

"What are the differences in safety and efficacy between auxiliary liver transplantation utilizing small-for-size grafts and conventional liver transplantation for the treatment of portal hypertension?"

ELIGIBILITY:
Inclusion Criteria:

1. Age > 14 years.
2. Presence of decompensated portal hypertension.
3. Meeting the indications for liver transplantation surgery.
4. International Normalized Ratio (INR) < 2.4.
5. Scheduled to undergo orthotopic auxiliary partial liver transplantation or conventional liver transplantation.

Exclusion Criteria:

1. Rare liver-related anatomical variations.
2. Presence of contraindications to liver transplantation combined with malignant tumors.
3. Grade III or higher portal vein thrombosis.
4. Severe systemic diseases unrelated to the etiology or complications of portal hypertension.
5. Special surgical procedures such as dual-graft liver transplantation.
6. Special graft sources including domino liver transplantation.
7. Liver re-transplantation.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cirrhotic portal hypertension who were treated at the Liver Transplantation Center of Beijing Friendship Hospital, Capital Medical University between January 2014 and December 2028, and who underwent either auxiliary liver transplantation using small-for-size grafts (study group) or conventional liver transplantation (control group).
Sampling Method: Non-Probability Sample
Enrollment: 396 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | Within one year after liver transplantation
Complications | Within one year after liver transplantation
portal hypertension resolution | Within one year after liver transplantation

IPD SHARING:
Plan to Share IPD: No